CLINICAL TRIAL: NCT01987570
Title: Effect of Allopurinol Administration on the Prevention of Muscle Mass Loss in Subject Immobilized.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALMU_2011; 2011-003541-17 (EudraCT Number)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2015-07

CONDITIONS: Patients With Grade II Ankle Sprain
Keywords: Xanthine oxidase; Magnetic resonance; Oxidative stress; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Experimental): One tablet of allopurinol is administrated orally at a dose of 300 mg/24 hours, during the time that the patient remains immobilized for 15 days.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): One tablet/24 hours of placebo orally, during the time that the patient remains immobilized for 15 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol
  Other Names: 1H-pirazolo (3,4-d)pirimidina-4-ol; Zyloric
  Arms: Allopurinol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Generating critical levels of power is a prerequisite for performing simple daily activities, such as rising from a chair or climbing stairs. For a young healthy person these activities can be performed easily, however after a prolonged period of forced inactivity (such as during the recovery from a sports injury, prolonged bed rest or spaceflight) a loss of muscle mass occurs. It has been suggested that this loss may be triggered by oxidative stress. An enzyme involved in the production of free radicals in various experimental models, including immobilization, is xanthine oxidase (XO). Although allopurinol is an inhibitor of XO widely used in clinical practice, its effect on the maintenance of muscle mass after an immobilization protocol is unknown. Thus, the major aim of this clinical trial is to determine the effect of allopurinol administration on the prevention of muscle mass loss in immobilized subjects.

This is a prospective, randomized study in which fifty young male subjects (aged between 25 and 40 years) diagnosed with grade II ankle sprain will be recruited. After immobilization the patients will be assigned randomly to one of two experimental groups, one treated with allopurinol (n=25) and the other with placebo (n=25). The dosage of allopurinol will be the same as recommended for gout patients, i.e. 300 mg/day orally, during all the immobilization period, which will last fifteen days. This medication will be delivered to the patients when they agree to participate in the clinical trial. They will be immobilized by posterior knee splint, preventing use of that leg.

We will determine muscle mass loss by performing two magnetic resonances of both legs before and after the immobilization period. We will also take two blood samples (before and after immobilization) to measure oxidative stress parameters (malondialdehyde, protein carbonyls, and XO activity), inflammatory parameters (IL-6, C-reactive protein and 1-antichymotrypsin), as well as vitamin D levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade II sprain.
* Boys
* Age 20-40 years.
* Patient without regular medication.
* All patients must provide written informed consent specific to this study complete.

Exclusion Criteria:

* Liver and gastrointestinal disease.
* Untreated hypothyroidism.
* Alcohol and / or drug addiction.
* Vitamin supplements.
* Eating Disorders.
* Drugs that decrease the concentration of lipids.
* Antihypertensive drugs.
* Athletes who exercise intensely.
* Mental disorders, depression or anxiety intensive. These conditions make the patient unable to understand the nature or the scope and possible consequences of the study.
* Patients presenting an infectious process and / or inflammatory before collecting the sample.
* Patients may not follow the protocol because of its lack of cooperation, to their inability to return to subsequent visits and there is little chance of completing the study procedures.
* Hypersensitivity to allopurinol

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2012-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Muscle mass loss | Day 0 and day 15
  Checks the loss of muscle mass percentage with Magnetic Resonance before and after treatment.
The role of xanthine oxidase in the loss of muscle mass | Day 0 and day 15
  Measure xanthine oxidase activity in plasma

SECONDARY OUTCOMES:
size of the leg muscles in a group of immobilized subjects. | Day 0 and day 15
  Checks the loss of muscle mass size with Magnetic Resonance before and after treatment.
oxidative stress parameters | Day 0 and day 15
  Glutathione (GSH), glutathione disulfide (GSSG), malondialdehyde (MDA) and oxidized proteins, after a period of immobilization of 15 days duration.

CONTACTS AND LOCATIONS:
Overall Officials: JOSÉ VIÑA, MD PhD (HON), Study Director — University of Valencia
Locations (2):
- Spain (2):
  - University of Valencia, Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia